CLINICAL TRIAL: NCT02962466
Title: Cumulus Cell Messenger Ribonucleic Acid (mRNA) Analysis as Oocyte Quality Marker in the Fertility Lab in a Prospective Multicenter Study
Brief Title: Multicenter Prospective Cumulus Cell Test Study
Acronym: MC_CC-Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BUN:143201628797
Record Dates: First submitted 2016-10-27; First posted 2016-11-11 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CC-Test diagnosis and Day 3 transfer (Experimental): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos + the extra cumulus cell based diagnosis and transfer of the best embryo based on morphology and CC diagnosis on day 3 of embryo growth (cleavage stage embryo).
  Interventions: Other: CC-Test
- D3 transfer control group (No Intervention): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on day 3 of embryo growth (cleavage stage embryo).
- D5 transfer control group (No Intervention): Patients undergo the standard ART treatment, as prescribed by the treating physician, with standard morphology based scoring of the embryos and transfer of the best embryo based on day 5 of embryo growth (blastocyst stage embryo).

INTERVENTIONS:
Other: CC-Test — classification of the oocyte based on the expression pattern observed in the cumulus cells
  Arms: CC-Test diagnosis and Day 3 transfer

SUMMARY:
Performing an additional non invasive oocyte diagnostic test based on cumulus gene expression could improve the outcome of the ART cycle.

DETAILED DESCRIPTION:
Background:

Currently, embryo selection before embryo transfer is done on the basis of morphological characteristics only. The morphology based selection procedure has only a limited predictive value. The need of an additional oocyte/embryo evaluating method is therefore required. This method should preferentially be: non invasive, objective, and available early in development. Each oocyte is surrounded with cumulus cells, cells which are normally disposed of during the assisted reproductive technique (ART)-procedure. A diagnostic test based on the cumulus cells fits al of the required criteria. In the current study the use of an oocyte diagnostic test based on cumulus cell gene expression is evaluated.

Primary purpose:

Validate a non invasive diagnostic test, not curing the infertility condition but improving the ART-treatment and as such reducing the physical and psychological effect of the (eventually failed) ART procedure or the potential side effects of this procedure on the patients.

Quality assurance plan for Data check and Source Data Verification:

The aim, the study design, the eligible patient population, the study plan and specific requirements were discussed on several occasions at the test sites. Clear collaborative agreements were made between the partners involved in this study. These stipulate the study protocol and the required action from each party at the specific time points and communication procedures. A trial initiation meeting was conducted on site by the PI. Interim evaluations for site monitoring and validation of data registration are foreseen. These will be initiated as soon as 10 patients are included in the study and can occur with every extra 5 patients being included. Data checks and verifications are foreseen on regular basis to be done by the trained study managers from the different study centers.

Definitions:

For study patients and matched controls serum human chorionic gonadotropin (hCG) is measured on day 14-17 after pick up. If positive, the hCG is followed up at day 20 and 25 (positive beta-hCG Pregnancy). All patients with a positive hCG are further followed up: 1) to detect a development of the foetal sac with positive heartbeat in weeks 7-8 of pregnancy (Clinical Pregnancy), 2) to have a routine ultrasound evaluation at weeks 12, 20 and 32 of pregnancy, 3) to have data on delivery and child health (Live Birth). The total number of pregnancies obtained from the stimulation cycles included in the study will be referred to as the Cumulative Pregnancy for each of the study groups.

Study design and Data analysis:

The study is a prospective matched control and assessor blind study. Most of the details on the study design are already described else ware in this document. It should however be noted that the assessor performing the additional diagnosis for the oocytes using the CC-Test is blind for eventual development of the oocyte into an embryo and the quality of these embryo based on the morphology.

Sample size was assessed based on retrospective studies performed by the Follicle Biology research laboratory (FOBI) UZBrussel. These indicated that with an ongoing pregnancy rate (OPR) in the two control groups of 30-40% and an expected OPR of 50%-70% the number of participants required is 20 to distinguish the difference with a power of 80%. For this reason at least 30 informative patients will be included in each study arm for each test site.

Clinical patient data related to the inclusion and exclusion criteria should be available and evaluated by the local investigator prior to enrolment of the patient in the study. Absence of any data related to the evaluation of the ART procedure or outcome will exclude this patient from further analysis. Data inconsistency or out of range results will be considered as absent data.

The statistical analysis of the results will be performed by a professional statistician experienced with the field, terminology and endpoints, using the best fit statistical method for each endpoint. For the analysis of the primary and secondary endpoints these include amongst others: Chi-square analysis, Kaplan-Meier analysis and multiple regression analysis, based on generalized linear models.

Interim analysis:

A first evaluation will be done when 20 cases, having had transfer after the CC-Test, are completed. This will comprise data on positive beta-hCG pregnancy, clinical pregnancy (7weeks).

ELIGIBILITY:
Inclusion Criteria:

* scheduled for intracytoplasmatic sperm injection (ICSI) and single embryo transfer on day 3
* patients down regulated with gonadotropin-releasing hormone (GnRH) antagonist and stimulated with Highly Purified human Menopausal Gonadotropin (HP-hMG)
* no more than 2 previous IVF or ICSI cycles with transfer prior to this one.
* Body mass index (BMI) should be higher than 17 and lower than 32
* patients should have regular menstrual cycles (between 24 and 35 days).

Exclusion Criteria:

* are smokers (>10 cigarettes per day)
* patients requesting Prenatal Genetic Diagnosis
* patients having polycystic ovary syndrome (PCOS), or Severe Endometriosis (AFS Stage 3-4)
* couples where the partner has an extremely low sperm count e.g.: extreme oligo-astheno-teratozoospermia (OAT), (<100.000/ml) or testicular sperm extraction (TESE)
* results of eventual preceding cycles may not indicate a known genetic disease, or low ovarian response or an oocyte maturation defect.

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy as observed by ultrasound | 2 months after embryo transfer
  this observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database

SECONDARY OUTCOMES:
positive beta-hCG Pregnancy as observed by serum analysis | 12-17 days after transfer
  this observation is routinely performed by the treating physician for every patient undergoing standard ART treatment and is thus available from the fertility center database
Live Birth by questionaire | et least 9 months after embryo transfer
  this observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database
Cumulative Pregnancy | 2 years after pick up
  this is the compilation of the data gathered in endpoint 1 and 3 for eventual consecutive cycles. This observation is routinely performed by the study nurses of the fertility center for every patient undergoing standard ART treatment and is thus available from the fertility center database.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Adriaenssens, Msc, Principal Investigator — Universitair Ziekenhuis Brussel; Johan Smitz, Prof. Dr., Study Director — Universitair Ziekenhuis Brussel
Locations (2):
- Belgium (2):
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - ULB Erasme, Anderlecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Van Vaerenbergh I, Adriaenssens T, Coucke W, Van Landuyt L, Verheyen G, De Brucker M, Camus M, Platteau P, De Vos M, Van Hecke E, Rosenthal A, Smitz J. Improved clinical outcomes after non-invasive oocyte selection and Day 3 eSET in ICSI patients. Reprod Biol Endocrinol. 2021 Feb 19;19(1):26. doi: 10.1186/s12958-021-00704-5. PMID 33608027